CLINICAL TRIAL: NCT05460871
Title: Evaluating the Efficacy and Safety of Pregabalin in Total Knee Arthroplasty Patients With Central Sensitization
Brief Title: Pregabalin for Central Sensitization in TKA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment lower than anticipated; none of the subjects completing the study.
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Lee A. Kral, Clinical Assistant Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202105361
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Osteo Arthritis Knee; Central Nervous System Sensitization
Keywords: Arthroplasty; Pain; Central Nervous System Sensitization; Osteo Arthritis Knee; Pregabalin
MeSH Terms: conditions — Pain | interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: Open label interventional trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Participants will receive standard peri-operative pain management
- Study (Pregabalin) (Experimental): Participants will receive pregabalin orally 75mg twice daily x 7 days prior to surgery, 150mg twice daily x 7 days after surgery, followed by 75mg twice daily x 7 days. Then Stop.
  Interventions: Drug: Pregabalin 75mg

INTERVENTIONS:
Drug: Pregabalin 75mg — participants will receive pregabalin orally 75mg twice daily x 7 days prior to surgery, then 150mg twice daily x 7 days after surgery, followed by 75mg twice daily x 7 days, then stop.
  Other Names: Study
  Arms: Study (Pregabalin)

SUMMARY:
The study purpose is to determine if giving pregabalin before and after total knee arthroplasty (TKA) can improve pain and meaningful function after surgery in patients that have central sensitization (CS).

Participants will be identified who are indicated for TKA. Interested patients will complete a standard Knee Injury and Osteoarthritis Outcomes Score (KOOS), asked their pain score (on a scale of 0 to 10), and complete the Central Sensitization Inventory (CSI). If they meet inclusion criteria and agree to participate, they will complete the informed consent before being randomized 1:1 to usual care (control group) or pregabalin (study group). The study group participants will take pregabalin starting 7 days prior to surgery. They will also be scheduled to have a pre-operative physical therapy (PT) appointment which will include tests and measures standard to PT. Tests will include a Timed Up and Go Test (TUG), a Sit to Stand 5 Times Repeat Test (5TSTS) and Patient Specific Functional Scale (SFS) measures.

On the day of surgery participants will be asked about any adverse effects of study medication and determine need to withdraw from study. The post-operative plan will be reviewed, including dose of study medication. For the pregabalin group the doses will be doubled for 7 days, then reduced for 7 days, then off. All participants will be given standard peri-operative pain management for TKA . All participants will complete standard of practice physical therapy.

After surgery (usually within 7 days) a physical therapist will perform standard post-operative evaluation and treatment for all participants. This includes a re-evaluation of the same pre-operative functional tests of TUG, 5TSTS and PSFS outcome measures. The study pharmacist will also call the patient to determine if there are any medication-related adverse effects and how much opioid medication the patient is taking at that time (morphine milligram equivalents- MME/day on average).

At the 6 week post-operative visit all participants will again complete the KOOS survey, report a pain score, complete the CSI survey and determine MME based on patient report of quantity of opioid medication used. A physical therapist will complete the functional assessment of the TUG, 5TSTS and PSFS outcome measures.

DETAILED DESCRIPTION:
The study purpose is to determine if giving pregabalin before and after total knee arthroplasty (TKA) can improve pain and meaningful function after surgery in patients that have central sensitization (CS). Central sensitization occurs when the brain (central nervous system) becomes hypersensitized and hypervigilant, over-reacting to any painful (and sometimes nonpainful) stimuli. Patients with greater central sensitization have been shown to have significantly more pain after surgery, including TKA. We are proposing to explore whether treatment with a nerve pain medication, pregabalin, can improve post-operative pain and function in these patients. This medication has been shown to improve central sensitization pain in the chronic pain setting but has not been studied for this purpose in the acute surgical pain setting.

Participants will be identified at the visit in which they are indicated for TKA. Patients indicated for a TKA will be approached about participating in the study. Either at that visit or later by phone or e-mail, interested patients will complete a standard Knee Injury and Osteoarthritis Outcomes Score (KOOS), which is part of the standard orthopedic evaluation. They will also be asked their pain score (on a scale of 0 to 10), and complete the Central Sensitization Inventory (CSI). If they meet study inclusion criteria, and they agree to participate, they will complete the informed consent (in person or on-line) and then be randomized 1:1 to usual care (control group) or pregabalin (study group). The study group participants will take pregabalin starting 7 days prior to surgery. The participant will receive usual medication counseling for this medication. They will also be scheduled to have a pre-operative physical therapy (PT) appointment at the time of their pre-op visit, which will include tests and measures standard to PT, but must include a Timed Up and Go Test (TUG), a Sit to Stand 5 Times Repeat Test (5TSTS) and Patient Specific Functional Scale (SFS) measures.

On the day of surgery participants will be asked about any adverse effects of study medication, and determine need to withdraw from study (for any reason). The post-operative plan will also be reviewed, including dose of study medication, for the pregabalin group. For the pregabalin group the doses will be doubled for 7 days, then reduced for 7 days, then off. All participants will be given standard peri-operative pain management for TKA (a nerve block and/or spinal unless contraindicated, anti-inflammatory drugs (NSAID) and acetaminophen (unless contraindicated) as well as oral opioid (usually oxycodone or hydromorphone) to use as needed for severe pain. All participants will complete standard of practice physical therapy on day of surgery or until discharged to home.

After surgery (usually within 7 days) a physical therapist will perform standard post-operative evaluation and treatment for all participants. This includes a re-evaluation of the same pre-operative functional tests of TUG, 5TSTS and PSFS outcome measures. At this time, the pharmacist will also call the patient to determine if there are any medication-related adverse effects and how much opioid medication the patient is taking at that time (morphine milligram equivalents- MME/day on average).

Standard follow-up after TKA is 6 weeks. At this visit all participants will again complete the KOOS survey, report a pain score, complete the CSI survey and determine, based on patient report, of quantity of opioid medication used (MME). A physical therapist will complete the functional assessment of the TUG, 5TSTS and PSFS outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing native joint unilateral TKA due to Grade 3-4 primary osteoarthritis
* Patients with score of at least 40 on Central Sensitization Inventory
* Patients who will complete PT within the U of Iowa Health Care system
* Patients who have been nonsmokers for > 2 years
* Patients between the ages of 50 and 85

Exclusion Criteria:

* Patients already taking pregabalin or had an adverse effect with pregabalin in the past
* Patients indicated for joint revision surgery
* Patients taking at least 30 morphine milligram equivalents per day for the past 1 month
* Patients with an estimate GFR < 30 ml/min
* Patients who do not have an understanding of English
* Patients who are pregnant or women of child-bearing years
* Patients who are prisoners
* Patients who score < 40 on the CSI
* Patients who answer Yes to any questions on the Columbia Suicide Severity Rating Scale or express suicidal ideation

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Kral, Pharm. D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After participants signed their informed consent, the participants completed surveys (Columbia Suicide Severity Rating Screen and Central Sensitization Inventory) to determine if they met the study inclusion criteria. Due to the sensitive nature of these surveys, our local IRB required that informed consent be signed before completing the assessments. If suicidal or the participant did not demonstrate Central Sensitization, they were not eligible for continued participation.
Period: Overall Study
Arm/Group | Control | Study (Pregabalin)
Started | 1 | 2
Completed | 0 | 0
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Study (Pregabalin) | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (0) | 55.5 (4.5) | 57.6 (4.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3
Grade 3-4 primary osteoarthritis [Count of Participants; unit: Participants] | 1 | 2 | 3
no previous adverse reaction to study drug [Count of Participants; unit: Participants] | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Calculate the Change Using the Knee Osteoarthritis Outcome Survey- Activities of Daily Living Subscale
Description: The difference in change on the Knee Osteoarthritis Outcome Survey (KOOS) - Activities of Daily Living subscale will be calculated between the treatment groups. The survey will be administered at baseline and at the subject's 6-weeks post procedure follow-up. The survey is scored on a continuous scale as follows: 1 = none, 2 = mild, 3 = moderate, 4 = severe, 5 = extreme.
Time Frame: Approximately 6 weeks
Population: No subjects completed baseline or follow-up surveys.
Arm/Group | Control | Study (Pregabalin)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Calculate the Change Using the Knee Osteoarthritis Outcome Survey-Symptoms
Description: The difference in change on the Knee Osteoarthritis Outcome Survey (KOOS) - Symptoms subscale will be calculated between the treatment groups. The survey will be administered at baseline and at the subject's 6-weeks post procedure follow-up. The survey is scored on a continuous scale as follows: 1 = never, 2 = rarely, 3 = sometimes, 4 = often, 5=always.
Time Frame: Approximately 6 weeks
Population: No subjects completed both the baseline and follow-up survey.
Arm/Group | Control | Study (Pregabalin)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Calculate the Change Using the Knee Osteoarthritis Outcome Survey-Stiffness
Description: The difference in change on the Knee Osteoarthritis Outcome Survey (KOOS) - Stiffness subscale will be calculated between the treatment groups. The survey will be administered at baseline and at the subject's 6-weeks post procedure follow-up. The survey is scored on a continuous scale as follows: 1 = none, 2 = mild, 3 = moderate, 4 = severe, 5 = extreme.
Time Frame: Approximately 6 weeks
Population: No subjects completed both the baseline and follow-up survey.
Arm/Group | Control | Study (Pregabalin)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Calculate the Change Using the Knee Osteoarthritis Outcome Survey-Sports and Recreational Activities
Description: The difference in change on the Knee Osteoarthritis Outcome Survey (KOOS) - Sports and Recreational Activities subscale will be calculated between the treatment groups. The survey will be administered at baseline and at the subject's 6-weeks post procedure follow-up. The survey is scored on a continuous scale as follows: 1 = none, 2 = mild, 3 = moderate, 4 = severe, 5 = extreme.
Time Frame: Approximately 6 weeks
Population: No subjects completed both the baseline and follow-up survey.
Arm/Group | Control | Study (Pregabalin)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Calculate the Change in Central Sensitization Inventory Score
Description: The difference in change on the Central Sensitization Inventory assessment will be calculated between the treatment groups. The survey will be administered at baseline and at the subject's 6-weeks follow-up. The survey is scored on a continuous scale as follows: 1 = never, 2 = rarely, 3 = sometimes, 4 = often, 5 = always.
Time Frame: Approximately 6 weeks
Population: No subjects completed both the baseline and follow-up survey.
Arm/Group | Control | Study (Pregabalin)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Calculate the Change of Physical Function Using the Timed Up & Go Assessment
Description: The change of physical function using the Timed Up & Go Assessment (TUG) will be evaluated at four intervals during the study; baseline, during the immediate post-operative time period (day of surgery or post-operative day 1), 7-day follow-up, and at 6-week follow-up. Patients will stand up from a chair, walk approximately 10 feet, turn, walk back and sit back down. This activity will be timed in seconds. The change from baseline until 6-week follow-up will be reported.
Time Frame: Approximately 6 weeks
Population: No subjects completed both the baseline and follow-up assessment.
Arm/Group | Control | Study (Pregabalin)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Calculate the Change of Physical Function Using the Stand to Sit Assessment
Description: The change of physical function using the Stand to Sit Assessment (STS) will be evaluated at four intervals during the study; baseline, during the immediate post-operative time period (day of surgery or post-operative day 1), 7-day follow-up, and at 6-week follow-up. Patients will stand up and sit down from a chair 5 times in a row, as quickly as they can. This activity will be timed in seconds. The change from baseline until 6-week follow-up will be reported.
Time Frame: Approximately 6 weeks
Population: No subjects completed both the baseline and follow-up assessment
Arm/Group | Control | Study (Pregabalin)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Calculate the Change of Physical Function Using the Patient-Specific Functional Scale Assessment
Description: The change of physical function using the Patient-Specific Functional Scale Assessment (PSFS) will be evaluated at four intervals during the study; baseline, during the immediate post-operative time period (day of surgery or post-operative day 1), 7-day follow-up, and at 6-week follow-up. At baseline, patients will asked to identify activities they are having difficulty/unable to do and would like to gain the mobility back after procedure. The activities will be scored on a continuous rating with The change from baseline until 6-week follow-up will be reported.
Time Frame: Approximately 6 weeks
Population: No subjects completed both the baseline and follow-up assessment
Arm/Group | Control | Study (Pregabalin)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Measure the Amount of Pain Reported After Procedure
Description: Using a numerical rating scale (0-10), patients will be asked to report their pain level. The scale is from 0 to 10 with 0 being no pain and 10 representing the most intense pain. The pain scores will be collected on 7-day post procedure follow-up and at the 6-week follow up. The change between the timepoints will be reported.
Time Frame: Approximately 6 weeks
Population: No subjects completed both the baseline and follow-up measurements
Arm/Group | Control | Study (Pregabalin)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Measure Post-operative Opioid Usage
Description: Review with subjects the type and amount of additional pain (opioid) medication required to control their pain. This will be examined approximately 7-day post procedure and at the 6-week post procedure follow-up. The amount of opioid medication taken by the subject will be converted to morphine equivalents for reporting purposes.
Time Frame: Approximately 6 weeks
Population: No subjects completed this.
Arm/Group | Control | Study (Pregabalin)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 3 months
Arm/Group | Control | Study (Pregabalin)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT05460871/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT05460871/ICF_001.pdf